CLINICAL TRIAL: NCT05474664
Title: Phase 2 Open-label, Single-arm, Multi-center Clinical Trial to Evaluate the Efficacy and Safety of Camostat Mesylate in Patients with Protein-losing Enteropathy After Fontan Operation
Brief Title: Camostat Mesylate for Protein-losing Enteropathy After Fontan Operation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Gi Beom Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FontanPLE
Record Dates: First submitted 2022-07-23; First posted 2022-07-26 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-10

CONDITIONS: Fontan Operation; Protein-Losing Enteropathy; Camostat Mesylate
Keywords: Fontan operation; Protein-Losing Enteropathy; Camostat mesylate
MeSH Terms: conditions — Protein-Losing Enteropathies | interventions — camostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- protein-losing enteropathy after Fontan operation (Experimental): single-arm with protein-losing enteropathy after Fontan operation
  Interventions: Drug: Camostat mesylate

INTERVENTIONS:
Drug: Camostat mesylate — 1. 4~12 years old: Camostate mesylate 100 mg, 2 times a day
  2. greater than 13 years old: Camostate mesylate 100 mg, 3 times a day

SUMMARY:
This study is phase 2 open-label, single-arm, multi-center clinical trial to evaluate the efficacy and safety of Camostat mesylate in patients with Protein-losing enteropathy after Fontan operation.

ELIGIBILITY:
Inclusion Criteria:

* history of protein-losing enteropathy after Fontan operation

  * more than 6 months after Fontan operation
  * more than 3 months of protein-losing enteropathy history (ascites, edema, diarrhea, etc) and less than 3.0 mg/dL of serum albumin without evidence of renal or liver disease

Exclusion Criteria:

* inability to take oral camostate mesylate
* hypersensitivity to camostate mesylate
* patients with taking similar medication or prohibited combination drug
* patients participating in other clinical trials
* patients with diet limitation
* patients with genetic disease such as galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Serum albumin | 6 months
  change compared with baseline

SECONDARY OUTCOMES:
Serum albumin | 6 months
  change ratio compared with baseline
Stool alpha-1 antitrypsin | 6 months
  change compared with baseline
Stool alpha-1 antitrypsin | 6 months
  change ratio compared with baseline
diarrhea | 6 months
  change of presence and number
ascites | 6 months
  ascites amount change by abdominal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Gi Beom B Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Daehak-ro Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park WY, Kim GB, Lee SY, Baek JS, Kim SJ, Jung J, Hyun MC, Lim YT, Lee H, Ko H, Lee J. Phase 2 Open-label, Single-arm, Multi-center Clinical Trial to Evaluate the Efficacy and Safety of Camostat Mesylate in Patients with Protein-losing Enteropathy After Fontan Operation. Pediatr Cardiol. 2025 Apr 14. doi: 10.1007/s00246-025-03859-9. Online ahead of print. PMID 40227431